CLINICAL TRIAL: NCT03244995
Title: An Online Dyadic Mind-Body Intervention for Glioma Patients and Their Partners
Brief Title: Mind-Body Intervention in Glioma Couples
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0290; NCI-2018-01099 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0290 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; Low Grade Glioma; Malignant Glioma; Metastatic Malignant Neoplasm in the Brain; Partner; WHO Grade III Glioma
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — Mind-Body Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (CBMB program) (Experimental): Patients undergo CBMB program consisting of 4-5 deep-breathing and meditation exercise sessions over 60 minutes and 2 weekly telephone calls over 15 minutes for 6 weeks. Patients also complete questionnaires regarding health, mood, sleeping habits, relationship, health care, work productivity, and quality of life.
  Interventions: Procedure: Mind-Body Intervention Procedure; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (waitlist control) (Active Comparator): Patients complete questionnaires as in Group I. Patients may undergo CBMB program after completion of study.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Mind-Body Intervention Procedure — Undergo CBMB program
  Other Names: Mind-Body Interventions; Mind-Body Medicine
  Arms: Group I (CBMB program)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well a couple-based mind body program works in improving spiritual, psychosocial, and physical quality of life in patients with high or low grade glioma or tumors that have spread to the brain and their partners. A couple-based mind body program may help to improve spiritual well-being, sleep difficulties, depressive symptoms, and overall quality of life in patients with glioma or tumors that have spread to the brain and their partners.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the feasibility of the couple-based mind-body (CBMB) program in patients with high grade glioma (HGG) and their partners.

II. Establish the initial efficacy of the CBMB program in patients and their partners regarding spiritual (primary), psychological and physical quality of life (QOL) (secondary) outcomes relative to a waitlist control (WLC) group.

EXPLORATORY OBJECTIVES:

I. Explore potential mediation (i.e., mindfulness, compassion, holding back, and intimacy) and moderation (e.g., baseline medical, demographic and psychosocial factors) effects of the intervention.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (CBMB PROGRAM): Patients undergo CBMB program consisting of 4-5 deep-breathing and meditation exercise sessions over 60 minutes and 2 weekly telephone calls over 15 minutes for 6 weeks. Patients also complete questionnaires regarding health, mood, sleeping habits, relationship, health care, work productivity, and quality of life.

GROUP II (WAITLIST CONTROL): Patients complete questionnaires as in Group I. Patients may undergo CBMB program after completion of study.

After completion of study, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT ONLY: Patients with a diagnosis of HGG or low grade glioma (LGG), based on radiographic or pathologic diagnosis of grade III or IV listed in the medical records, or patients with a malignancy that has metastasized to the brain
* PATIENT ONLY: Patients must be within 1 month of initiating or having undergone any type of cancer treatment (i.e., surgery, radiotherapy, chemotherapy)
* PATIENT ONLY: Karnofsky performance status (KPS) of 80 or above
* PATIENT ONLY: Having a spouse/romantic partner (including same-sex) and who is willing to participate
* PATIENT & PARTNER: Able to read and speak English
* PATIENT & PARTNER: Able to provide informed consent
* PATIENT & PARTNER: Have access to internet connectivity

Exclusion Criteria:

* PATIENT ONLY: Regularly (self-defined) participation in psychotherapy or a formal cancer support group
* PATIENT ONLY: Cognitive deficits that would impede the completion of self-report instruments as deemed by the clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-08-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of couple-based mind-body program (CBMB) as determined by overall accrual | Up to 6 weeks
  Trial considered feasible if 50% of eligible couples consent. Will calculate rates, frequencies, and 90% confidence intervals (CIs), as applicable.
Feasibility of CBMB program as determined by attrition | Up to 6 weeks
  Trial considered feasible if 80% of enrolled couples complete T1 and T2 assessments. Will calculate rates, frequencies, and 90% CIs, as applicable.
Feasibility of CBMB program as determined by adherence | Up to 6 weeks
  Trial considered feasible if 50% of all sessions are attended. Will calculate rates, frequencies, and 90% CIs, as applicable.
Feasibility of CBMB program as determined by acceptability | Up to 6 weeks
  Trial considered feasible if > 75% of patients in the CBMB group rate the intervention as acceptable. Will calculate rates, frequencies, and 90% CIs, as applicable.
CBMB program efficacy | Up to 6 weeks
  Will calculate effect sizes for pairwise between-group comparisons of intervention outcomes at T2. Will test for between-group differences in the change of scores between T1 and T2 using analysis of variance.

OTHER OUTCOMES:
CBMB program efficacy on quality of life (QOL) outcomes | Up to 3 months after completion of study
  Will examine treatment mediators and moderators. Will examine if treatment efficacy on QOL outcomes measured at T3 is potentially achieved through improved mindfulness, self-compassion, holding back and intimacy measured at T2 using linear regression analysis in both a and b paths. Ninety percent bootstrap CIs will be constructed to assess the significance of the indirect effects defined using the product-of-coefficient approach. Linear regression analysis or multi-level modeling will be used to test for the interaction effects between treatment and baseline mindfulness, self-compassion, holding back and intimacy, as well as baseline medical and demographic factors (i.e., sex, age, and Karnofsky performance status), each at a two-sided significance level of 0.1.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org